CLINICAL TRIAL: NCT02250118
Title: Phase I Study to Determine the Maximum Tolerated Dose and Evaluate the Pharmacokinetics of Intrapleural Bevacizumab After Pleural Drainage in Patients With Symptomatic Malignant Pleural Effusion in the Context of Breast Cancer
Brief Title: Intrapleural Bevacizumab After Pleural Drainage in the Context of Breast Cancer
Acronym: BEVAP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: Institut Curie (Other)
Collaborators: Henri Mondor University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2014-02; 2014-000654-11 (EudraCT Number)
Record Dates: First submitted 2014-09-08; First posted 2014-09-26 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-05

CONDITIONS: Pleural Effusion, Malignant; Breast Cancer
Keywords: pleural; effusion; breast; cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Breast Neoplasms; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Intrapleural use: range 0.5 - 5 mg/kg
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Intrapleural Bevacizumab
  Other Names: Avastin

SUMMARY:
Metastatic pleural effusion is a common complication of late-stage cancer and reduces the quality of life and survival of patients. The survival of patients with recurrent pleurisy by uncontrolled local or systemic treatment is less than 6 months. It is important to develop specific therapies to improve the quality of life and survival of patients with metastatic pleurisy.

Bevacizumab is a monoclonal anti vascular endothelial growth factor (VEGF) which has proven effective in many indications in oncology. Vascular endothelial growth factor (VEGF) is an angiogenic factor which increases endothelial permeability. It plays a central role in many tumors of epithelial origin. In this context, it is legitimate to ask whether an antiangiogenic targeting VEGF may be effective in patients with metastatic pleurisy by decreasing local blood supply and over-permeability.

No study has been interested in the intra-pleural pharmacokinetics of monoclonal antibodies and there are no predictive or prognostic biomarkers for metastatic pleural effusions.

The investigators believe that intrapleural administration of bevacizumab will reduce the pleural vasculature permeability. It will neutralize VEGF present in pleural fluid and reduce the replenishment of effusion due to its prolonged half-life of 21 days.

The investigators therefore propose a phase I study to determine the maximum tolerated dose and the recommended dose for phases II, studying the pharmacokinetics of intrapleural bevacizumab administered by an implantable device after evacuating a symptomatic metastatic pleurisy as part of a mammary carcinoma. The VEGF intrapleural levels and serum will be study and the time until a new puncture. Dyspnea will be evaluated as well as its impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically documented pleural effusion in a type of breast carcinoma in exudate or with no other identified cause. In the absence of positive cytology, will ensure that there is no other cause of the patient's history may explain the effusion.
2. Unilateral or bilateral malignant pleural effusion but requiring drainage on only one side.
3. Patient presenting an indication for pleural implantable device, means that requiring at least one pleural drainage.
4. Patient aged 18 years old or more and without measure of legal protection
5. Subject female or male
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
7. Expected life span > 2 months
8. Corticosteroids authorized if started less than 15 days before enrollment and no dose modification will be allowed during treatment
9. Adequate biological functions 14 days before inclusion:

   * Haemoglobin ≥ 8 g/dl (transfusion authorized)
   * Neutrophil count (ANC) ≥ 1000/mm3
   * Platelet count ≥ 100 000/mm3
   * International Normalized Ratio (INR) ≤ 1.5 and/or Prothrombin Ratio (TR) ≥ 70 % and Partial Thromboplastin Time (PTT) ≤ 1.5
   * Aspartate Aminotransferase Test (AST), Alanine Aminotransferase Test (ALT), Gamma-Glutamyl Transpeptidase (GGT), Alk Phos ≤ 3 times Unit Line Number (ULN), bilirubin ≤ 40 μmol/L
   * Lactate Dehydrogenase (LDH) ≤ 1,5 times ULN
   * Albumin ≥ 28 g/dL
   * Creatinine clearance ≥ 45 mL/min according to the Modification of the Diet in Renal Disease formula (MDRD)
   * Proteinuria ≤ 1g/dL in the absence of tract infection
10. Cardiac Function satisfactory: Left Ventricular Ejection Fraction (LVEF) determined by myocardial scintigraphy or echocardiography
11. Females of childbearing potential must take acceptable methods of birth control during the complete duration of treatment and serum pregnancy tests must be negative at the inclusion. Men must agree to use a condom if his partner is of child bearing potential
12. Patient receiving a social security system
13. Signed inform consent

Exclusion Criteria:

1. Pregnant or lactating women or childbearing potential refusing methods of birth control
2. Transudative pleural effusion: pleural protein < 30 g/L and/or Light's criteria when pleural protein is not indicative. Light's criteria are as follows (for diagnosis of transudative):

   * Pleural protein/serum protein ratio < 0.5
   * Pleural LDH/serum LDH ratio < 0.6
   * Pleural LDH < two-thirds the upper limit of normal of serum LDH
3. Purulent pleural effusion.
4. Macroscopically haemorrhagic pleural effusion.
5. Bilateral metastasis pleurisy requiring punctures on both sides.
6. Any co morbidity considered to be incompatible with participation in the study, according to the investigator, particularly: untreated infectious disease, chronic respiratory insufficiency, chronic renal insufficiency, Child Pugh B or C, hepatocellular insufficiency; chronic heart failure not controlled by appropriate medical treatment.
7. Contraindications to intrapleural administration of bevacizumab:

   * Non-controlled arterial or venous thromboembolism
   * Major surgery during the previous month or planned after study
   * Known, non treated brain metastases
   * Known hypersensitivity to bevacizumab or one of its excipients
   * Hypersensitivity to Chinese hamster ovary cell (CHO) products or other human recombinant or humanized antibodies
   * Intravenous administration of bevacizumab planned or underway in the usual cancer treatment (≥ 3 weeks wash out from the intrapleural injection)
   * Radiotherapy including lung field concerned since the administration of the product until the end of the study.
8. Diagnosis of any second malignancy within the last 5 years, except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for > 3 years.
9. Patients can't participate in another clinical trial with another experimental anti-cancer drug therapy simultaneously for 90 days. No exclusion period is required after the end of the trial visit.
10. Impossibility to follow the calendar of exams because of geographic, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | 90 days after intrapleural injection
  Maximum tolerated dose (MTD) according to safety of intrapleural bevacizumab at dose levels of 1 mg/kg, 3 mg/kg and 5 mg/kg administered by pleural catheter after drainage of symptomatic malignant pleural effusion in a context of breast cancer.

SECONDARY OUTCOMES:
Study of the pleural and serum pharmacokinetics | 90 days
  Pharmacokinetics of bevacizumab just before administration and 1 hour after treatment on Day 1, and at D15, D30, D60 and D90.
Study of pleural and serum Vascular Endothelial Growth Factor (VEGF) levels | 90 days
  Pleural and serum VEGF levels just before administration and 1 hour after treatment on Day 1, and at D15, D30, D60 and D90.
Determination of time until new punction or death | 2 years
  Response to treatment assessed by the time to new puncture
Total number of pleural drainage procedures | 90 days
  Measure of the total number of pleural drainage procedures at D15, D30, D60 and D90.
Drainage-free survival and overall survival | 2 years
  Drainage-free survival and overall survival Evaluation of survival without punction and overall survival
Evaluation of dyspnoea | 90 days
  Measure by dyspnoea scale and peak flow at D15, D30, D60 and D90
Evaluation of quality of life | 2 years
  Quality of life (QLQ-C30) questionnaire according to European Organisation for Research and Treatment of Cancer (EORTC) and FACIT questionnaire Dyspnoea 10 Short Form at D15, D30, D60 and D90 and every 6 month during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maya Gutierrez, MD, Principal Investigator — Institut Curie - Hôpital René Huguenin
Locations (1):
- Institut Curie - Hôpital René Huguenin, Saint-Cloud, France